CLINICAL TRIAL: NCT03952884
Title: Skeletal Muscle Protein Synthetic Response to Amino Acid and Peptides
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Nicholas Burd, Assistant Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 18897
Record Dates: First submitted 2019-05-08; First posted 2019-05-16 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Protein Metabolism
Keywords: Metabolism; Amino Acid Peptides; Muscle Protein Synthesis; Muscle Protein Breakdown
MeSH Terms: interventions — Resistance Training; Leucine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Leucine (Active Comparator): Participants will be allocated to an exercise or non-exercise group. After resistance exercise (or equivalent time point for non-exercise group), participants will consume 2g leucine powder dissolved in 250 mL of water.
  Interventions: Behavioral: Resistance Exercise; Behavioral: No Resistance Exercise; Dietary Supplement: Leucine
- Leucine Peptide (Dileucine) (Experimental): Participants will be allocated to an exercise or non-exercise group. After resistance exercise (or equivalent time point for non-exercise group), participants will consume 2g protein peptide powder dissolved in 250 mL of water.
  Interventions: Behavioral: Resistance Exercise; Behavioral: No Resistance Exercise; Dietary Supplement: Dileucine

INTERVENTIONS:
Behavioral: Resistance Exercise — Prior to protein consumption participants will perform an acute bout of resistance exercise. They will warm up with two sets of 10 repetitions at 35-75% working load respectively, then perform four working sets of 10-12 repetitions at 65-70% of 1-RM. 1 min, 30 sec rest periods will be implemented between each set.
Behavioral: No Resistance Exercise — Participants allocated to this group will not perform exercise prior to the administration of the nutritional intervention. Participants will remain at rest throughout the trial.
Dietary Supplement: Leucine — Participants will be given 2g of leucine dissolved in 250mL of water. Drink will be consumed immediately after exercise or equivalent time point for non-exercise group.
  Arms: Leucine
Dietary Supplement: Dileucine — Participants will be given 2g of dileucine dissolved in 250mL of water. Drink will be consumed immediately after exercise or equivalent time point for non-exercise group.
  Arms: Leucine Peptide (Dileucine)

SUMMARY:
Skeletal muscle quality is an important determinant of exercise performance and overall health. It is vital for not just movement, but also metabolizing nutrients. Protein from the diet can promote muscle protein synthesis for muscle recovery and growth. More importantly, doing so shifts net protein balance positively (e.g. protein synthesis is greater than protein breakdown) and promotes greater rates of muscle protein turnover. Leucine is an amino acid required to build muscle, but it also acts as a signaling molecule informing the muscle to start protein synthesis. Before reaching skeletal muscle, dietary protein is digested into small peptides and free amino acids. Rate of absorption from the intestine to the blood stream is significantly faster for peptides compared to amino acids. As amino acid availability in the blood is a precursor for muscle protein synthesis, our objective is to determine if the different absorption rates between free amino acid and peptides influence muscle protein synthetic and breakdown rates.

ELIGIBILITY:
Inclusion Criteria:

* Recreationally-active adults: ≥ 30 min of physical activity at moderate intensity ≥ 3 times per week
* Ages: 18-35 years old
* English fluency

Exclusion Criteria:

* Tobacco, nicotine (patch/gum) use (previous 6 mo)
* Alcohol consumption >10 drinks per week
* Metabolic disorders (e.g., Metabolic Syndrome, Diabetes, thyroid diseases)
* Cardiovascular disease, arrhythmias
* Hypogonadism
* Asthma
* History of uncontrolled hypertension
* Orthopedic injury/surgery (within 1 yr)
* Hepatorenal, musculoskeletal, autoimmune, or neurological disease
* History of neuromuscular problems
* Previous participation in amino acid tracer studies
* Predisposition to hypertrophic scarring or keloid formation
* Consumption of ergogenic-levels of dietary supplements that may affect muscle mass (e.g., creatine, HMB), insulin-like substances, or anabolic/catabolic pro-hormones (e.g., DHEA) within 6 weeks prior to participation
* Consumption of thyroid, androgenic, or other medications known to affect endocrine function
* Consumption of medications known to affect protein metabolism (e.g., prescription-strength corticosteroids, non-steroidal anti-inflammatories, or acne medication)
* Currently pregnant

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-05-03 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-11-20 (Actual)

PRIMARY OUTCOMES:
Fractional Synthetic Rate of Mixed Muscle Proteins | Postabsorptive for 3.5 hours, Postprandial for 3 hours.
  Mixed muscle protein synthesis rates will be assessed during the 3.5hr Postabsorptive period (e.g. non-fed state) and the 3hr postprandial period (e.g. fed state) for both experimental interventions (e.g. leucine and leucine peptide). This will allow us to assess the change in fractional synthetic rate from the Postabsorptive period to the postprandial period.
Fractional Synthetic Rate of Myofibrillar Proteins | Postabsorptive for 3.5 hours, Postprandial for 3 hours.
  Myofibrillar muscle protein synthesis rates will be assessed during the 3.5hr Postabsorptive period (e.g. non-fed state) and the 3hr postprandial period (e.g. fed state) for both experimental interventions (e.g. leucine and leucine peptide). This will allow us to assess the change in fractional synthetic rate from the Postabsorptive period to the postprandial period.
Fractional Breakdown Rate of Mixed Muscle Proteins | Postprandial for 1 hour
  Mixed muscle protein breakdown rates will be assessed during the first hour of the postprandial period (e.g. fed state) for both experimental interventions (e.g. leucine and leucine peptide). This will allow us to assess the change in fractional breakdown rate for each respective experimental intervention.

SECONDARY OUTCOMES:
Phosphorylation of muscle anabolic signaling | Baseline, immediately after ingestion of leucine/leucine peptides, and 3 hours after ingestion of leucine/leucine peptides
  Phosphorylation of anabolic signaling pathways will be assessed in the fasted state and after the ingestion of the experimental interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas A. Burd, Ph.D., Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- Freer Hall, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2019-06-20): https://cdn.clinicaltrials.gov/large-docs/84/NCT03952884/ICF_000.pdf